CLINICAL TRIAL: NCT01938963
Title: The Depression/Hypertension in Chinese Older Adults-Collaboration in Health
Brief Title: Chinese Older Adults-Collaboration in Health (COACH)Study
Acronym: COACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Zhejiang University (Other); University of Pennsylvania (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Yeates Conwell, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH100298-01 (NIH)
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Depression; Hypertension
Keywords: Depression; Hypertension; Older Adults
MeSH Terms: conditions — Depression; Hypertension | interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Care as usual (No Intervention)
- Collaborations in Health (COACH) (Experimental): COACH integrates the care provided by the older person's primary care provider (PCP) with that delivered by an Aging Worker (AW; a lay member of the village's Aging Association), supervised by a psychiatrist consultant. Based on chronic disease management principles, the PCP is trained to use evidence based practice guidelines for treatment of both HTN and depression, and provided with access to mental health consultation regarding optimal management of the patient's depression. The AW is trained to conduct a systematic assessment of the older person's social context to identify and reduce social and environmental barriers to treatment adherence and response. AWs participate with the PCP in developing multi-disciplinary care plans for their shared patients, reinforce treatment adherence and adoption of healthy behaviors, and emphasize activation and engagement of the older person in activities designed to improve their connectedness to others and to the community.
  Interventions: Behavioral: Collaborations in Health (COACH)

INTERVENTIONS:
Behavioral: Collaborations in Health (COACH) — Primary care provider, aging worker, and Psychiatrist Consultant are trained to collaborate in their shared clients' care.
  Arms: Collaborations in Health (COACH)

SUMMARY:
This study will see if education of village doctors and aging workers in identification and management of hypertension and depression, using standardized procedures,consultation with a psychiatrist as needed, and collaborations between the village doctor and aging worker in care elderly patients in the village better achieve better outcomes for their depression and high blood pressure than usual care.

DETAILED DESCRIPTION:
The Depression/Hypertension in Chinese Older Adults - Collaborations in Health (COACH) Study is a randomized controlled trial (RCT) comparing the COACH intervention to care as usual (CAU) for the treatment of comorbid depression and hypertension (HTN) in Chinese older adult rural village residents. COACH integrates the care provided by the older person's primary care provider (PCP) with that delivered by an Aging Worker (AW; a lay member of the village's Aging Association), supervised by a psychiatrist consultant. Based on chronic disease management principles, the PCP is trained to use evidence based practice guidelines for treatment of both HTN and depression, and provided with access to mental health consultation regarding optimal management of the patient's depression. The AW is trained to conduct a systematic assessment of the older person's social context to identify and reduce social and environmental barriers to treatment adherence and response. AWs participate with the PCP in developing multidisciplinary care plans for their shared patients, reinforce treatment adherence and adoption of healthy behaviors, and emphasize activation and engagement of the older person in activities designed to improve their connectedness to others and to the community. Finally, PCP, AW, and Psychiatrist Consultant are trained to collaborate in their shared clients' care.

One hundred and sixty villages will be randomized to deliver COACH or CAU to eligible subjects who reside there (approximately 15 per village will meet criteria), or a total of about 2400 subjects. Treatment will continue for one year, with research evaluations at baseline, 3 6, 9, and 12 months.

Specific aims of the study are to determine whether COACH is more effective than CAU in treating depression (Aim 1) and HTN (Aim 2); whether improvements in treatment adherence precede reductions in depression and improvement in BP control (Aim 3a), and whether improvements in depression symptoms precede improvements in BP control (Aim 3b); if COACH is associated with greater improvements in health related quality of life than CAU (Aim 4); and to compare the costs associated with each approach (Aim 5).

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling residents registered to the selected village, and thus also registered patients of the village's PCP.
* Age ≥ 60 years, the typical retirement age in rural China.
* Clinically significant depression defined as baseline PHQ-9 score ≥ 10.
* Diagnosis of hypertension
* Intact cognitive functioning (6-Item Screener score <3) to assure ability to participate with the treatment team in management of their conditions.
* Capable of independent communication
* Capacity to give informed consent.

Exclusion Criteria:

* Incapable (no capacity) of giving verbal consent to this study.
* Acute high suicide risk at baseline assessment. Patients assessed to be dangerously suicidal at later assessments will be discontinued from the study, their providers notified, and their safety guaranteed.
* Psychosis, alcoholism. We exclude patients with psychosis or active alcoholism in the past 6 months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2685 (Actual)
Dates: Start 2014-01; Primary Completion 2018-02-09 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
Depressive symptom change | baseline, 3-, 6-, and 12-month follow up
  The measure for depressive symptom change will be the Hamilton Depression Rating Scale.

SECONDARY OUTCOMES:
Adherence to antidepressant and antihypertensive medication recommendations | baseline, 3-, 6-, 9-, and 12-month follow up
  First, the Morisky Medication Adherence Measure will be used. Secondly, a Medication Possession Ratio will be used-a combination of pill counts and verification of pharmacy refills.

OTHER OUTCOMES:
Hypertension | baseline, 3-, 6-, 9-, and 12-month follow-up
  Blood pressure readings will be taken at baseline and at follow-ups.
Health related quality of life | baseline, 3-, 6-, 9-, and 12-month follow up
  Quality of life will be measured using the World Health Organization Quality of Life- short version, WHOQOL-BREF.
  Satisfaction will be measured with the Client Satisfaction Questionnaire 8-item.
Costs associated with the intervention | baseline, 3-, 6-, 9-, and 12-month follow-up
  Two components will be evaluated: program costs associated with adding resources to care as usual, and medical costs attributed to the care of the subjects in each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Yeates Conwell, MD, Principal Investigator — University of Rochester; Shulin Chen, MD, PhD, Principal Investigator — Zhejiang University, Department of Psychology
Locations (7):
- United States (4):
  - Tulane University, New Orleans, Louisiana
  - Regents of the University of Michigan, Ann Arbor, Michigan
  - University of Rochester Medical Center, Rochester, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
- China (3):
  - Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Provincial Committee on Aging, Hangzhou
  - Zhejiang Provincial Center for Disease Control and Prevention, Hangzhou

REFERENCES:
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Derived] Chen S, Conwell Y, Xue J, Li L, Zhao T, Tang W, Bogner H, Dong H. Effectiveness of integrated care for older adults with depression and hypertension in rural China: A cluster randomized controlled trial. PLoS Med. 2022 Oct 24;19(10):e1004019. doi: 10.1371/journal.pmed.1004019. eCollection 2022 Oct. PMID 36279299
- [Derived] Chen S, Conwell Y, Xue J, Li LW, Tang W, Bogner HR, Dong H. Protocol of an ongoing randomized controlled trial of care management for comorbid depression and hypertension: the Chinese Older Adult Collaborations in Health (COACH) study. BMC Geriatr. 2018 May 29;18(1):124. doi: 10.1186/s12877-018-0808-1. PMID 29843644